CLINICAL TRIAL: NCT02738294
Title: Necessity Assessment of Magnifying Endoscopy With Narrow Band Imaging Targeted Biopsy Compared With Endoscopic Forceps Biopsy From White Light Endoscopy
Brief Title: Necessity Assessment of ME-NBI Targeted Biopsy Compared With EFB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, MD.Ph.D, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: rjxhnk[2013]113
Record Dates: First submitted 2016-03-08; First posted 2016-04-14 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2016-03

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Suspected EGC group (Experimental): Participants with suspected EGC from white light endoscopy were enrolled.The endoscopist first used white light endoscopy to identify suspected gastric lesions and assessed lesions carefully with magnifying view, non-magnifying NBI view and ME-NBI view in sequence. After assessing suspected EGC in ME-NBI view, ME-NBI targeted biopsy was performed where abnormal phenomenon was identified in ME-NBI view.
  Interventions: Device: ME-NBI observation and ME-NBI targeted biopsy

INTERVENTIONS:
Device: ME-NBI observation and ME-NBI targeted biopsy — The endoscopist assessed lesions which were suspected EGC carefully with ME-NBI. After assessing suspected EGC in ME-NBI view, ME-NBI targeted biopsy was performed where abnormal phenomenon was identified in ME-NBI view.

SUMMARY:
The aim of the present study was to assess whether it was necessary to conduct magnifying endoscopy with narrow band imaging (ME-NBI) targeted biopsy compared with endoscopic forceps biopsy (EFB) from white light endoscopy in diagnosing early gastric cancer (EGC). Meanwhile, the investigators proposed the most cost-effective way to diagnose EGC.

DETAILED DESCRIPTION:
ME-NBI has been widely used for the diagnosis of stomach diseases, especially in the early diagnosis of gastric cancer. The aim of the present study was to evaluate diagnostic efficacy of ME-NBI targeted biopsy and ME-NBI combined with targeted biopsy compared with EFB from white light endoscopy and ME-NBI combined with EFB.

A prospective study was conducted encompassing suspected EGC. All patients were performed white light endoscopic examination with EFB and then ME-NBI with ME-NBI targeted biopsy. Outcome measures were assessed and compared, including diagnostic efficacy of EFB from white light endoscopy,ME-NBI combined with EFB, ME-NBI targeted biopsy and ME-NBI combined with targeted biopsy.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients with gastric lesions detected by white light endoscopy and suspected of EGC

Exclusion Criteria:

* they had advanced gastric cancer
* lesions were histopathologically confirmed to be submucosal tumors
* they had a history of gastrectomy
* tissue biopsy wasn't obtained or more than 2 biopsies were performed on suspected gastric lesions during last white light endoscopy
* they couldn't tolerate another endoscopic examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Accuracy in distinguishing high-grade neoplasia (HGN) from non-HGN | 30 months
  EFB and ME-NBI targeted biopsy and final resected specimens were assessed according to the Vienna classification. Suspected lesions were assessed in ME-NBI view according to the diagnostic classification proposed by Yao and Ezoe et al. However, little different from their classification, lesions were classified into positive HGN phenomenon, indefinite and suspected HGN, negative HGN phenomenon. After that, ME-NBI targeted biopsy was performed where abnormal or suspected phenomenon was observed. Compared with final pathology of endoscopic submucosal dissection (ESD) or surgery specimens, sensitivity of EFB, ME-NBI, ME-NBI targeted biopsy, ME-NBI combined EFB and ME-NBI combined targeted biopsy was calculated. Accuracy of EFB and ME-NBI targeted biopsy was compared using McNemar test. The same method was used to compare ME-NBI combined EFB and ME-NBI combined targeted biopsy.
Sensitivity in distinguishing HGN from non-HGN | 30 months
  EFB and ME-NBI targeted biopsy and final resected specimens were assessed according to the Vienna classification. Suspected lesions were assessed in ME-NBI view according to the diagnostic classification proposed by Yao and Ezoe et al. However, little different from their classification, lesions were classified into positive HGN phenomenon, indefinite and suspected HGN, negative HGN phenomenon. The former classification was diagnosed as HGN. The latter two classification was diagnosed as HGN. After that, ME-NBI targeted biopsy was performed where abnormal or suspected phenomenon was observed. Compared with final pathology of ESD or surgery specimens, sensitivity of EFB, ME-NBI, ME-NBI targeted biopsy, ME-NBI combined EFB and ME-NBI combined targeted biopsy was calculated. Sensitivity of EFB and ME-NBI targeted biopsy was compared using McNemar test. The same method was used to compare ME-NBI combined EFB and ME-NBI combined targeted biopsy.
Specificity in distinguishing HGN from non-HGN | 30 months
  EFB and ME-NBI targeted biopsy and final resected specimens were assessed according to the Vienna classification. Suspected lesions were assessed in ME-NBI view according to the diagnostic classification proposed by Yao and Ezoe et al. However, little different from their classification, lesions were classified into positive HGN phenomenon, indefinite and suspected HGN, negative HGN phenomenon. The former classification was diagnosed as HGN. The latter two classification was diagnosed as HGN. After that, ME-NBI targeted biopsy was performed where abnormal or suspected phenomenon was observed. Compared with final pathology of ESD or surgery specimens, specificity of EFB, ME-NBI, ME-NBI targeted biopsy, ME-NBI combined EFB and ME-NBI combined targeted biopsy was calculated. Specificity of EFB and ME-NBI targeted biopsy was compared using McNemar test. The same method was used to compare ME-NBI combined EFB and ME-NBI combined targeted biopsy.

SECONDARY OUTCOMES:
Positive predictive value (PPV) in distinguishing HGN from non-HGN | 30 months
  EFB and ME-NBI targeted biopsy and final resected specimens were assessed according to the Vienna classification. Suspected lesions were assessed in ME-NBI view according to the diagnostic classification proposed by Yao and Ezoe et al. However, little different from their classification, lesions were classified into positive HGN phenomenon, indefinite and suspected HGN, negative HGN phenomenon. The former classification was diagnosed as HGN. The latter two classification was diagnosed as HGN. After that, ME-NBI targeted biopsy was performed where abnormal or suspected phenomenon was observed. Compared with final pathology of ESD or surgery specimens, PPV of EFB, ME-NBI, ME-NBI targeted biopsy, ME-NBI combined EFB and ME-NBI combined targeted biopsy was calculated.
Negative predictive value (NPV) in distinguishing HGN from non-HGN | 30 months
  EFB and ME-NBI targeted biopsy and final resected specimens were assessed according to the Vienna classification. Suspected lesions were assessed in ME-NBI view according to the diagnostic classification proposed by Yao and Ezoe et al. However, little different from their classification, lesions were classified into positive HGN phenomenon, indefinite and suspected HGN, negative HGN phenomenon. The former classification was diagnosed as HGN. The latter two classification was diagnosed as HGN. After that, ME-NBI targeted biopsy was performed where abnormal or suspected phenomenon was observed. Compared with final pathology of ESD or surgery specimens, NPV of EFB, ME-NBI, ME-NBI targeted biopsy, ME-NBI combined EFB and ME-NBI combined targeted biopsy was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Gastroenterology and Clinical Laboratory, Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided